CLINICAL TRIAL: NCT06232876
Title: Continuous Versus Intermittent Ward Monitoring on Vital Sign Abnormalities, Clinical Interventions, and Serious Complications: the CONSTANT Trial
Brief Title: Continuous Versus Intermittent Ward Monitoring
Acronym: CONSTANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, Daniel Sessler, Professor and Vice President for Clinical and Outcomes Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSC-MS-24-0978
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blinded continuous vital sign monitoring (Sham Comparator): Continuous ward monitoring with vital signs recorded but not available to patients, clinicians, or investigators.
  Interventions: Device: Blinded continuous vital sign monitoring
- Unblinded continuous vital sign monitoring (Experimental): Continuous ward monitoring with vital signs available to clinicians and investigators.
  Interventions: Device: Unblinded continuous vital sign monitoring

INTERVENTIONS:
Device: Blinded continuous vital sign monitoring — Continuous ward monitoring with vital signs recorded but not available to patients, clinicians, or investigators.
  Arms: Blinded continuous vital sign monitoring
Device: Unblinded continuous vital sign monitoring — Continuous ward monitoring with vital signs available to clinicians and investigators.
  Arms: Unblinded continuous vital sign monitoring

SUMMARY:
The investigators will randomize adults having major non-cardiac inpatient surgery to blinded versus unblinded continuous postoperative vital sign monitoring (saturation, ventilation, and heart rate). The investigators will use a wearable, untethered, and battery-powered sensor (Masimo Radius PPG, Masimo, Irvine, CA) that wirelessly connects to a Masimo monitor and continuously records saturation, ventilation, and pulse rate.

The primary outcome will be areas-exceeding-thresholds for desaturation (<85%), bradypnea (<7 breaths/min), tachypnea (>30 breaths/min), tachycardia (heart rate >130 beats/min), and bradycardia (heart rate <45 beats/min). These exposure thresholds represent a balance between events that are clinically meaningful and excessive alarms that will discourage clinician participation. The investigators expect about 2 alerts per patient per day with these thresholds, with most being considered informative or actionable by nurses. In unblinded patients, clinician alerts will be activated at these thresholds.

DETAILED DESCRIPTION:
Postoperative cardiovascular mortality remains common, and a third occurs during the initial hospitalization. Deterioration occurs over many hours but is usually unrecognized because vital signs are evaluated a 4-6-hour intervals, just as they were a half-century ago when patient acuity was much lower. Recognition of even subtle changes in basic vital signs may allow clinicians to detect cardiopulmonary deterioration well before serious adverse events occur. Consequent clinical interventions may in turn prevent complications, or at least moderate their severity. The investigators therefore propose a single-center randomized trial of continuous ward monitoring.

The investigators will randomize adults having major non-cardiac inpatient surgery to blinded versus unblinded continuous vital sign monitoring (saturation, ventilation, and heart rate) and hourly intermittent blood Postoperative cardiovascular mortality remains common, and a third occurs during the initial hospitalization. Deterioration occurs over many hours but is usually unrecognized because vital signs are evaluated 4-6-hour intervals, just as they were a half-century ago when patient acuity was much lower. Recognition of even subtle changes in basic vital signs may allow clinicians to detect cardiopulmonary deterioration well before serious adverse events occur. Consequent clinical interventions may in turn prevent complications, or at least moderate their severity. The investigators therefore propose a single-center randomized trial of continuous ward monitoring.

The Investigators will randomize adults having major non-cardiac inpatient surgery to blinded versus unblinded continuous postoperative vital sign monitoring (saturation, ventilation, and heart rate). The investigators will use a wearable, untethered, and battery-powered sensor (Masimo Radius PPG, Masimo, Irvine, CA) that wirelessly connects to a Masimo monitor and continuously records saturation, ventilation, and pulse rate.

The primary outcome will be areas-exceeding-thresholds for desaturation (<85%), bradypnea (<7 breaths/min), tachypnea (>30 breaths/min), tachycardia (heart rate >130 beats/min), and bradycardia (heart rate <45 beats/min). These exposure thresholds represent a balance between events that are clinically meaningful and excessive alarms that will discourage clinician participation. The investigators expect about 2 alerts per patient per day with these thresholds, with most being considered informative or actionable by nurses. In unblinded patients, clinician alerts will be activated at these thresholds.

Secondarily, the investigators will evaluate a composite of clinical interventions for desaturation, bradypnea, tachypnea, tachycardia, and bradycardia. On an exploratory basis, as a pilot for a future major multi-center outcome trial, The investigators will evaluate a composite of major complications within 30 days after non-cardiac inpatient surgery including rapid response team activation, unplanned intubation, myocardial injury after non-cardiac surgery (MINS), non-fatal cardiac arrest, stroke, sepsis, in-hospital mortality, and hospital readmission.

The innovative long-term goal is to reduce in-hospital postoperative cardiovascular and pulmonary mortality. Specifically, The investigators expect to show that continuous rather than intermittent postoperative vital sign monitoring identifies unstable patients which will allow clinicians to intervene and prevent serious complications and death - thus promoting longer and healthier lives.

ELIGIBILITY:
Inclusion Criteria:

1. Are admitted to one of the wards equipped with the Masimo Radius PPG solution;
2. Are ≥18 years old;
3. Are designated American Society of Anesthesiologists physical status 1-4;
4. Had major noncardiac surgery lasting at least 1.5 hours;
5. Are expected to remain hospitalized at least two postoperative nights;
6. Had general anesthesia with or without neuraxial anesthesia.

Exclusion Criteria:

1. Have language, vision, or hearing impairments that may compromise continuous monitoring;
2. Are designated Do Not Resuscitate, hospice, or receiving end of life care;
3. Have previously participated in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Vital sign abnormalities with routine hospital monitors | 48 postoperative hours
  Area of vital sign abnormalities exceeding defined thresholds.

SECONDARY OUTCOMES:
Interventions | 48 postoperative hours
  The incidence of a composite of clinical interventions for desaturation, hypoventilation, tachypnea, tachycardia, bradycardia, and hypotension within 48 hours after major non-cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No